CLINICAL TRIAL: NCT06968481
Title: A Phase 2, Single-center, Open-label, Randomized, Dose Ascending Trial to Evaluate the Efficacy and Safety of Sublingual Oxytocin for the Prevention of Post-partum Hemorrhage Caused by Uterine Atony in Term Pregnant Women Having an Uncomplicated Vaginal Delivery
Brief Title: Sublingual Oxytocin for the Prevention of Post-partum Hemorrhage
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EX005-201
Record Dates: First submitted 2025-04-01; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Post Partum Hemorrhage
Keywords: sublingual oxytocin; oxytocin; post-partum hemorrhage; severe post-partum hemorrhage; SPPH; Prevention of post-partum hemorrhage; Efficacy and safety
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual Oxytocin (Experimental)
  Interventions: Drug: Oxytocin
- Intramuscular Oxytocin (Other): Reference product
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Sublingual oxytocin 1000 IU, 3000 IU or 6000 IU
  Arms: Sublingual Oxytocin
Drug: Oxytocin — Intramuscular oxytocin 10 IU
  Arms: Intramuscular Oxytocin

SUMMARY:
An open-label, randomized, single-center, dose ascending trial will be conducted to evaluate the efficacy and safety of sublingual oxytocin for the prevention of post-partum hemorrhage caused by uterine atony in term pregnant women having an uncomplicated vaginal delivery. The primary objective is to estimate the optimal effective dose (ED90) of sublingual oxytocin administered during the active management of the third stage of labor to result in satisfactory uterine tone and a cumulative blood loss < 500 ml at 20 minutes after vaginal delivery in 90% of parturients with an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Women willing and able to provide Informed consent.
2. Women who are able to understand, confirm and give informed consent during an antenatal visit or first stage of labor (cervical dilation <6 cm).
3. Healthy, primiparous or multiparous (2-4 deliveries), term-pregnant female with a gestational age of 37 to 42 weeks (inclusive). Gestational age should be confirmed with an obstetrical ultrasound if available.
4. Aged between 18 and 40 years (both inclusive).
5. Confirmed singleton pregnancy.
6. Based on the Investigator assessment, maternal and fetal conditions are met to expect a vaginal delivery.
7. For participants in the PK subgroup: women with baseline hemoglobin level ≥11 g/dL.

Exclusion Criteria:

1. Women who are unable to provide written Informed consent.
2. Women undergoing an elective or emergency cesarean section.
3. Conditions predisposing to uterine atony and PPH (e.g., previous PPH, placenta praevia, multiple gestation, severe pre-eclampsia, polyhydramnios, uterine fibroids, need for induction of labor, bleeding diathesis, sepsis, body mass index [BMI] ˃ 30 kg/m2 , macrosomia with estimated fetal weight >4500 g, if antenatal ultrasound was performed).
4. Women with moderate or severe anemia (defined as Hb <10 g/dL).
5. Women who have undergone female genital mutilation.
6. Known allergies to carbetocin, other oxytocin homologues or excipients in the medicinal products used in the trial.
7. Oral conditions before administration of sublingual oxytocin such as moderate erythema and edema, severe irritation/inflammation, moderate or severe abrasion.
8. Conditions predisposing to myocardial ischemia due to pre-existing cardiovascular diseases (such as hypertrophic cardiomyopathy, valvular heart disease and/or ischemic heart disease, including vasospasm of the coronary arteries) or known long QT syndrome or related symptoms.
9. Any clinically significant abnormality following review of medical history, laboratory result and physical examination at screening as judged by the Investigator (e.g., severe anemia, antepartum hemorrhage, mental disorder, history of cervical cancer or history of severe infection of the uterus, religious beliefs prohibiting blood transfusions).
10. Previous surgery of the cervix or uterus or any other preexisting condition that could interfere with the measurement of uterine contractility.
11. Current use or use within 30 days before the start of the IMP or reference product of one or more of predefined medications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 330 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a satisfactory uterine tone and cumulative blood loss < 500 ml | From administration of the drug to 20 minutes post-partum

SECONDARY OUTCOMES:
Proportion of participants with satisfactory uterine tone | after 3 min, 5 min, 10 min, 15 min, 30 min, 1 hour, 2 hours, 4 hours, 12 hours and 24 hours after administration of the drug
Measurement of blood loss | 3 min, 5 min, 10 min, 15 min, 30 min, 1 hour, 2 hours, 4 hours, 12 hours and 24 hours after administration of the drug
Proportion of participants who develop primary PPH | Up to 24 hours after administration of the drug
Incidence of blood transfusion due to PPH | At 24 hours after administration of the drug
Incidence of laparotomy for the treatment of PPH | At 24 hours after administration of the drug
Proportion of participants that achieve cessation of active bleeding | Within 20 minutes after administration of the drug
Time to PPH onset | Immediately after the intervention up to 24 hours post intervention
Time to active bleeding cessation | Immediately after the intervention up to 24 hours post intervention
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the time of written informed consent until the End of Study visit and must be followed up until resolution or stabilization
Absolute number and percentage of participants with oral irritation/inflammation and abrasion | after admission to hospital (during the Latent or Active phase for all participants) and at 20 minutes and 24 hours post dose for participants who are administered the investigational drug

CONTACTS AND LOCATIONS:
Locations (1):
- Africa Center of Excellence for Population Health and Policy, Kano, Kano State, Nigeria